CLINICAL TRIAL: NCT03401736
Title: A Study on the Relationship Between Biodiversity of Intestinal Microbiota in Patients and Different Sedative-hypnotics Undergoing Mechanical Ventilation
Brief Title: The Diversity of Intestinal Microbiota in Patients With Different Sedative-hypnotics Undergoing Mechanical Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Can't get enough participant
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, PI, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-443-T339
Record Dates: First submitted 2017-12-16; First posted 2018-01-17 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Intestinal Microbiota; Mechanical Ventilation
Keywords: Sedatives and Hypnotics
MeSH Terms: interventions — Respiration, Artificial; Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M：received midazolam (Experimental): Patients who requires the mechanical ventilation allocated to the midazolam group (group M) were treated with an infusion bolus of 0.05 mg/kg and continuous infusion of 0.04 to 0.20 mg/kg/hour, with the dosage adjusted to achieve the desired level of sedation.
  Interventions: Device: Mechanical Ventilation; Drug: Midazolam
- Group D: received dexmedetomidine (Active Comparator): Patients who requires the mechanical ventilation allocated to the dexmedetomidine group (group D) received an infusion bolus of 1 ug/kg within 10 minutes and continuous infusion of 0.25 to 0.75 ug/kg/hour, with the dosage adjusted to achieve the desired level of sedation.All patients maintained BIS between 65~85 and the Ramsay score was 3 to 4.
  Interventions: Device: Mechanical Ventilation; Drug: Dexmedetomidine

INTERVENTIONS:
Device: Mechanical Ventilation — Whether midazolam and dexmedetomidine have an effect on the diversity of intestinal microbiota or not is still unknown，especially the patient who requires the mechanical ventilation.
Drug: Midazolam — The impact of Midazolam on the diversity of intestinal microbiota.
  Other Names: Midazolam injection
  Arms: Group M：received midazolam
Drug: Dexmedetomidine — The impact of dexmedetomidine on the diversity of intestinal microbiota.
  Other Names: Dexmedetomidine injection
  Arms: Group D: received dexmedetomidine

SUMMARY:
Bidirectional communication between the CNS and the GI tract - the brain-gut axis - occurs both in health and disease.Patients with mechanical ventilation in ICU (ICU) often meet the necessary nutritional needs. These patients often appear varying degrees of intestinal flora imbalance, such as diarrhea, vomiting, abdominal distension and other complications, which exert negative effect on treatment and prolong hospitalization time.So far，whether the sedative drugs used for a long time in mechanically ventilated patients will affect the diversity of intestinal flora or not has not been reported.The effects of different sedative drugs on the intestinal flora diversity need further study.Therefore, this topic will used midazolam and dexmedetomidine to study the effect on the diversity of intestinal microbiota.Meanwhile，the research will provide a theoretical basis for rational use of mechanical ventilation and sedative drugs.

DETAILED DESCRIPTION:
There are a variety of normal microbial communities in the healthy human intestines, which maintain the physiological balance of the host. Under normal circumstances, there are about 104 intestinal microflora in the adult's intestines. The total number of genes is about 150 times the number of human genes. More and more studies have found that intestinal flora plays an important role in the occurrence of many human diseases. In recent years, the role of intestinal microflora in the brain axis has gradually been recognized and become a hot spot of research, and a new concept of the brain - gut axis is proposed.

The brain-gut axis is a bidirectional communication system between the central nervous system (CNS) and the gastrointestinal tract. Compared with ordinary mice, mild exposure to pressure can increase the level of corticosterone and adrenocorticotropic hormone in sterile mice, and this overreaction can be reversed by transplantation of normal rats' feces.Together, it is clear that the gut microbiota can be a key regulator of mood, cognition, pain, and obesity. Understanding microbiota-brain interactions is an exciting area of research which may contribute new insights into individual variations in cognition, personality, mood, sleep, and eating behavior.The abnormal expression of GABA (GABA) receptor in central nervous system is related to anxiety and depression. It is found that probiotics can regulate the expression of GABA receptor in the cerebral cortex through vagus nerve, thereby reducing anxiety and depression.5-HT signal system abnormalities may be associated with the pathophysiological changes of irritable bowel syndrome (IBS), while intestinal flora can affect the generation of neurotransmitter 5-HT in the intestine, resulting in changing of gastrointestinal motility and sensibility of internal organ. The above study means that the brain axis plays an important role in maintaining the diversity of intestinal microbiota.

It is essential that using sedatives to maintain the safety and comfort of the patient in ICU.Most patients also need receiving mechanical ventilation.Many patients in Intensive care unit appear varying degrees of intestinal microflora imbalance,especially received mechanical ventilation.So far,whether sedatives used for a long time in mechanically ventilated patients will affect the diversity of intestinal flora or not still not been reported. The effects of different sedative drugs on the intestinal flora diversity also need further study.Therefore, the topic will discuss the diversity of intestinal microbiota in patients with different sedative-hypnotics and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive long-term (≥12 hours) mechanical ventilation after operation on admission to the ICU
* APACHEII score 12-20 points
* no receive other clinical trials in the near 3 months
* no acute infectious disease, psychosis or other disease
* volunteer people

Exclusion Criteria:

* known or suspected allergy to midazolam or Dexmedetomidine
* suspected pregnancy, gross obesity, hyperlipemia, moribund state
* history of alcoholism or intake of anti-anxiety drugs or hypnotics
* chronic renal failure
* coma by cranial trauma or neurosurgery or unknown etiology or status epilepticus
* unwillingness to provide informed consent by patients or their authorized surrogates following ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The changing trends of the diversity of Intestinal microbiota | Up to 1 year from the beginning of the study
  Bacterial diversity revealed by 16S ribosomal RNA (rRNA) gene high-throughput sequencing (HTS).Feces were collected before operation from patients who had surgery.After the first collection, another was collected when the patient received mechanical ventilation more than 12 hours.

SECONDARY OUTCOMES:
The changing trends of weight | Up to 1 month from the beginning of the study
  The changing trends of weight was recorded in kilograms by the experimental assistant
duration of sedation | Time from achieving sedation until reaching full consciousness,up to 1 week.
  BIS and Ramsay score were described by the anesthetist physician
Duration of mechanical ventilation | Up to 3 days from the beginning of the study
  Duration of mechanical ventilation was described by the anesthetist physician

CONTACTS AND LOCATIONS:
Overall Officials: Li Jing Jie, M.D., Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai9 Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulak A, Bonaz B. Brain-gut-microbiota axis in Parkinson's disease. World J Gastroenterol. 2015 Oct 7;21(37):10609-20. doi: 10.3748/wjg.v21.i37.10609. PMID 26457021
- [Background] Evrensel A, Ceylan ME. Fecal Microbiota Transplantation and Its Usage in Neuropsychiatric Disorders. Clin Psychopharmacol Neurosci. 2016 Aug 31;14(3):231-7. doi: 10.9758/cpn.2016.14.3.231. PMID 27489376
- [Background] Al Omran Y, Aziz Q. The brain-gut axis in health and disease. Adv Exp Med Biol. 2014;817:135-53. doi: 10.1007/978-1-4939-0897-4_6. PMID 24997032
- [Background] Luna RA, Savidge TC, Williams KC. The Brain-Gut-Microbiome Axis: What Role Does It Play in Autism Spectrum Disorder? Curr Dev Disord Rep. 2016 Mar;3(1):75-81. doi: 10.1007/s40474-016-0077-7. Epub 2016 Feb 26. PMID 27398286
- [Background] Mayer EA, Padua D, Tillisch K. Altered brain-gut axis in autism: comorbidity or causative mechanisms? Bioessays. 2014 Oct;36(10):933-9. doi: 10.1002/bies.201400075. Epub 2014 Aug 22. PMID 25145752
- [Background] Li Q, Zhou JM. The microbiota-gut-brain axis and its potential therapeutic role in autism spectrum disorder. Neuroscience. 2016 Jun 2;324:131-9. doi: 10.1016/j.neuroscience.2016.03.013. Epub 2016 Mar 8. PMID 26964681
- [Background] van De Sande MM, van Buul VJ, Brouns FJ. Autism and nutrition: the role of the gut-brain axis. Nutr Res Rev. 2014 Dec;27(2):199-214. doi: 10.1017/S0954422414000110. Epub 2014 Jul 8. PMID 25004237
- [Background] Atkinson W, Lockhart S, Whorwell PJ, Keevil B, Houghton LA. Altered 5-hydroxytryptamine signaling in patients with constipation- and diarrhea-predominant irritable bowel syndrome. Gastroenterology. 2006 Jan;130(1):34-43. doi: 10.1053/j.gastro.2005.09.031. PMID 16401466
- [Background] Dizdar V, Spiller R, Singh G, Hanevik K, Gilja OH, El-Salhy M, Hausken T. Relative importance of abnormalities of CCK and 5-HT (serotonin) in Giardia-induced post-infectious irritable bowel syndrome and functional dyspepsia. Aliment Pharmacol Ther. 2010 Apr;31(8):883-91. doi: 10.1111/j.1365-2036.2010.04251.x. Epub 2010 Feb 2. PMID 20132151
- See also: Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial — https://www.ncbi.nlm.nih.gov/pubmed/?term=Dexmedetomidine+vs+midazolam+for+sedation+of+critically+ill+patients%3A+a+randomized+trial

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03401736/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03401736/ICF_001.pdf